CLINICAL TRIAL: NCT05963737
Title: PMI Guide PS Setting in Pressure Support-ventilated Patients - Prospective Multicenter Clinical RCT
Brief Title: PMI Guide PS Setting in Pressure Support-ventilated Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KY2023-005-02
Record Dates: First submitted 2023-07-01; First posted 2023-07-27 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-07

CONDITIONS: Mechanical Ventilation
Keywords: pressure support ventilation; inspiratory effort; inspiratory muscle pressure index

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm (Experimental): The initial PS level is set up based on VT/PBW (6-8ml/kg) and RR (20-30 breaths/min) when patients are enrolled in the experimental arm. The following steps need to be repeated every 2 hours for 48 hours. Step 1: 3 times short EIOs (2-3s) are performed. At least 1 minute between each occlusion. PMI is calculated as the mean value of 3 measured values. Step 2: Clarify whether PMI is in the target range (PMI 0-2cmH2O). If yes, keep this PS level. If not, implement step 3. Step 3: A downward or upward PS setting adjustment is performed at a 1cmH2O interval. Every PS level is maintained for 3-5 minutes. PMI is measured again and step 3 is repeated until the PMI target is reached. Step 4: supplemental adjustment: PS setting needs to be returned to the previous level if the patient presents the following signs: VT < 4 ml/Kg, RR > 35 breaths/min, respiratory acidosis, respiratory distress, VT > 10ml/Kg, Pplat > 30 cmH2O, respiratory alkalosis.
  Interventions: Procedure: PS setting strategy in pressure-support ventilated patients
- Control arm (No Intervention): Patients randomized to the control arm need to continue to accept the traditional ventilation strategy which is VT/PBW (6-8ml/kg) and RR (20-30breaths/min) guide PS setting.

INTERVENTIONS:
Procedure: PS setting strategy in pressure-support ventilated patients — Use PMI guide PS setting in pressure-supported ventilated patients and keep PMI within the target range (0-2cmH2O).
  Arms: Experimental arm

SUMMARY:
Pressure support ventilation (PSV) is an assistant mechanical ventilation mode, that is widely implemented in mechanical ventilation treatment but there are no exact guidelines to guide PS setting. Traditional PS setting strategy (VT/PBW 6-8ml/kg and RR 20-30 breaths/min)has risks of excessive or insufficient assistance. Inspiratory muscle pressure index (PMI) is a noninvasive respiratory mechanical indicator and is available at the bedside. PMI was correlated with inspiratory effort and has the potential ability to predict low inspiratory effort and high inspiratory effort. The primary objective of this study is to investigate the clinical validity of a PMI-guided PS setting strategy. Specifically, the investigators aim to evaluate its impact on inspiratory effort as well as its potential for lung and diaphragm protection. Additionally, the investigators seek to assess the effect of this ventilation strategy on mechanical ventilation outcomes while evaluating the feasibility of our trial protocol.

DETAILED DESCRIPTION:
Pressure support ventilation (PSV) is an assistant mechanical ventilation mode to provide synchronous inspiratory support for patients with spontaneous breathing and to efficiently reduce the workload imposed on the respiratory muscle. PSV is widely implemented in mechanical ventilation treatment but there are no exact guidelines to guide PS setting. Clinicians and respiratory therapists usually adjust ventilator parameters based on tidal volume/predicted body weight (VT/PBW, 6-8ml/kg) and current respiratory rate (RR, 20-30 breaths/min). This strategy has risks of excessive or insufficient assistance because the PS setting cannot be modulated dynamically based on the requirements of ventilated patients.

Inspiratory muscle pressure index (Pmus index, PMI) is defined as the difference between plateau pressure (Pplat) and airway peak pressure (Ppeak) during end-inspiratory occlusion (EIO). PMI is a noninvasive respiratory mechanical indicator and is available at the bedside like airway occlusion pressure (P0.1) because holding operations were integrated into the majority ventilator. Several studies showed PMI was correlated with inspiratory effort. Our previous study showed PMI has the potential ability to predict low inspiratory effort and high inspiratory effort, and the optimal cut-off PMI value was approximately 0 cmH2O and 2 cmH2O.

The primary objective of this study is to investigate the clinical validity of a PMI-guided PS setting strategy. Specifically, the investigators aim to evaluate its impact on inspiratory effort as well as its potential for lung and diaphragm protection. Additionally, the investigators seek to assess the effect of this ventilation strategy on mechanical ventilation outcomes while evaluating the feasibility of our trial protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients under PSV
* Predicted ventilated time of more than 48 hours.

Exclusion Criteria:

* Age less than 18 years old;
* Known pregnancy;
* BMI>35kg/m2;
* Brain-stem or cervical cord injury;
* Known or clinically suspected elevated intracranial pressure (ICP>18 mmHg);
* Nervus phrenicus or diaphragm injury;
* Broncho-pleural fistula;
* Chronic obstructive pulmonary disease (COPD);
* Pressure support ventilated time more than 48 hours before randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of conditions in the range of normal inspiratory effort per patient | up to 48 hours
  the time from the start of PSV mode to the successful weaning of the ventilated patients

SECONDARY OUTCOMES:
The duration of mechanical ventilation | up to 28 days
  the time from the start of mechanical ventilaion to the successful weaning of the patients
Tracheostomy rate | up to 28 days
  the proportion of all subjects who underwent tracheostomy
Reintubation rate | up to 28 days
  the proportion of all subjects who underwent reintubation
Diaphragm thickness (Tdi) | up to 28 days
  using the Tdi to estimate the change of diaphragm function and activity during PSV
Diaphragm thicken fraction (TFdi) | up to 28 days
  using the TFdi to estimate the change of diaphragm function and activity during PSV
Diaphragm excursion (EXdi) | up to 28 days
  using the EXdi to estimate the change of diaphragm function and activity during PSV
inspiratory muscle pressure (Pmus) | up to 28 days
  measuring Pmus to estimate the patient's inspiratory effort during the whole pressure-support ventilated duration
esophageal pressure time product (PTPes) | up to 28 days
  measuring PTPes to estimate the patient's inspiratory effort during the whole pressure-support ventilated duration
number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 28 days
  treatment-related adverse events including pneumothorax, circulatory instability, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao R, Yang YL, Zhang L, Miao MY, Zhou JX. Use of pressure muscle index to guide pressure support ventilation setting: a study protocol and statistical plan for a prospective randomised controlled proof-of-concept trial. BMJ Open. 2024 Aug 3;14(8):e082395. doi: 10.1136/bmjopen-2023-082395. PMID 39097307